CLINICAL TRIAL: NCT01482455
Title: Lipid-induced Insulin Resistance is Not Mediated by Impaired Transcapillary Transport of Insulin and Glucose in Humans
Brief Title: Fat and Transcapillary Insulin Transport
Acronym: FATRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FATRAIN
Record Dates: First submitted 2011-11-27; First posted 2011-11-30 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2012-09

CONDITIONS: Lipid-induced Insulin Resistance
Keywords: Insulin resistance; vascular impairment; diabetes
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Clamp/Glycerol (Placebo Comparator): Glycerol infusion (glycerol in 0.9% saline provided by the pharmacy of the Vienna General Hospital, will be applied at a rate of 0.7 mg.kg-1.min-1) in order to match the lipid-induced rise in serum glycerol concentrations in the same experimental setting. 0-240 min: Intralipid® 20%, Pharmacia AB, Stockholm, Sweden, 90 ml/hr; Heparin "Immuno"®, Immuno AG, Vienna, Austria, bolus: 200IU, continuous infusion: 0.2 IU.kg-1.min-1. After two hours, a hyperinsulinemic-euglycemic clamp (Actrapid, Novo Nordisk, Bagsvaerd, Denmark; 40 mU.m-2 body surface area min-1) test will be commenced (120-240 min).
  Interventions: Other: Elevation of FFA during Clamp
- OGTT/Lipid (Active Comparator): On study-day 1, four hours after start of a triglyceride/heparin infusion an oral glucose tolerance test (OGTT, 75g glucose dissolved in 300ml flavoured water) will be performed (240-420 min).
  Interventions: Other: Elevation of FFA during OGTT
- OGTT/Glycerol (Placebo Comparator): On study-day 2, four hours after start of a glycerol infusion an oral glucose tolerance test (OGTT, 75g glucose dissolved in 300ml flavoured water) will be performed (240-420 min).
  Interventions: Other: Elevation of FFA during OGTT
- Clamp/Lipid (Active Comparator): 0-240 min: Intralipid® 20%, Pharmacia AB, Stockholm, Sweden, 90 ml/hr; Heparin "Immuno"®, Immuno AG, Vienna, Austria, bolus: 200IU, continuous infusion: 0.2 IU.kg-1.min-1. After two hours, a hyperinsulinemic-euglycemic clamp (Actrapid, Novo Nordisk, Bagsvaerd, Denmark; 40 mU.m-2 body surface area min-1) test will be commenced (120-240 min).
  Interventions: Other: Elevation of FFA during Clamp

INTERVENTIONS:
Other: Elevation of FFA during OGTT — 0-240 min: Intralipid® 20%, Pharmacia AB, Stockholm, Sweden, 90 ml/hr; Heparin "Immuno"®, Immuno AG, Vienna, Austria, bolus: 200IU, continuous infusion: 0.2 IU.kg-1.min-1
  Arms: OGTT/Glycerol; OGTT/Lipid
Other: Elevation of FFA during Clamp — 0-240 min: Intralipid® 20%, Pharmacia AB, Stockholm, Sweden, 90 ml/hr; Heparin "Immuno"®, Immuno AG, Vienna, Austria, bolus: 200IU, continuous infusion: 0.2 IU.kg-1.min-1.
  Arms: Clamp/Glycerol; Clamp/Lipid

SUMMARY:
There is a current debate whether impaired insulin-mediated microvascular perfusion limits the delivery of hormones and nutrients to muscle and whether short term FFA elevation affects transcapillary transport of insulin and glucose thereby representing a rate-controlling step for insulin-stimulated muscular glucose disposal in humans.

To address these questions, the investigators determined the changes of interstitial glucose and insulin in skeletal muscle of healthy volunteers during intravenous administration of triglycerides or glycerol under physiologic and supraphysiologic hyperinsulinemic conditions.

DETAILED DESCRIPTION:
Increased lipid availability reduces insulin-stimulated glucose disposal in skeletal muscle, which is generally explained by lipid induced inhibition of myocellular insulin signalling, It remains unclear whether lipids also impair transcapillary transport of insulin and glucose which could thereby become rate-controlling for glucose disposal Increased accumulation and availability of lipids cause impaired skeletal muscle insulin sensitivity. It is yet unclear if transcapillary transport of insulin and glucose is impaired by acute elevation of free fatty acids and represents a rate-limiting step during the development of short-term lipid-induced insulin resistance. We determined the changes of interstitial glucose and insulin in skeletal muscle of healthy volunteers during intravenous administration of triglycerides and heparin or glycerol under physiologic and supraphysiologic hyperinsulinemic conditions.

ELIGIBILITY:
Inclusion Criteria:

* The volunteers have to be older than 19 years,
* nonobese (body mass index, BMI less than 27 kg/m2),
* normolipidemic (fasting serum concentration of triglycerides < 140 mg/dL and
* total cholesterol < 200 mg/dL) and
* non-smokers.

Exclusion Criteria:

* The following exclusion criteria will be applied:

  * any medication within two weeks prior to the start of study,
  * regular alcohol consumption > 40 g/d,
  * acute inflammatory disease defined by serum C-reactive protein > 1 mg/dL,
  * abnormalities in the screening visit or in laboratory tests considered as clinically relevant,
  * family history of diabetes mellitus or dyslipidemia,
  * glucose intolerance,
  * allergy or hypersensitivity against study medication,
  * blood clotting disorders.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Blood flow | between the start of the lipid/glycerol infusion until the end of the study (360 min)
  Regional blood flow. Muscular blood flow will be measured by the laser Doppler flow technique (LDF, Moor Instruments, Devon, UK) as described previously

SECONDARY OUTCOMES:
Interstitial insulin concentration | between the start of the lipid/glycerol infusion until the end of the study (360 min)
  Interstitial insulin concentration in skeletal muscle is measured via microdialysis based on sampling of analytes from the interstitial space fluid by means of a dialysis membrane at the tip of a microdialysis probe.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Principal Investigator — German Diabetes Center
Locations (1):
- Medical University Vienna, Vienna, Austria